CLINICAL TRIAL: NCT06684886
Title: Predictors of Diabetic Foot Outcome in Chronic Kidney Disease Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Eman Mahmoud Zaki Osman, resident doctor at nephrology department, Assiut University
Other Study IDs: diabetic foot CKD in patients
Record Dates: First submitted 2024-11-10; First posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Diabetic Foot Disease; Chronic Kidney Disease Due to Type 2 Diabetes Mellitus
Keywords: chronic kidney disease
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- diabetic foot group: diabetic nephropathy patients with diabetic foot
  Interventions: Other: Ankle Brachial Index
- non diabetic foot group: diabetic nephropathy patients without diabetic foot
  Interventions: Other: Ankle Brachial Index

INTERVENTIONS:
Other: Ankle Brachial Index — Normal ABI ranges from 1.0 - 1.4
  * Pressure is normally higher in the ankle than the arm.
  * Values above 1.4 suggest a noncompressible calcified vessel.
  * In diabetic or elderly patients, the limb vessels may be fibrotic or calcified. In this case, the vessel may be resistant to collapse by the blood pressure cuff, and a signal may be heard at high cuff pressures. The persistence of a signal at a high pressure in these individuals results in an artifactually elevated blood pressure value.
  * An value below 0.9 is considered diagnostic of PAD.
  * Values less than 0.5 suggests severe PAD.
  * Individuals with such severe disease may not have sufficient blood flow to heal a fracture or surgical wound; they should be considered for revascularization if they have a non-healing ulcer.

SUMMARY:
Individuals with diabetic neuropathy and Chronic kidney disease (CKD) are 15 times more likely to have a non-traumatic lower extremity amputation compared to those with DM alone . The incidence of DF and its evolution appear to be proportionally related to the stage of CKD . One of the most important causes is vascular calcification, which is common in patients with atherosclerosis, DM, CKD, and elderly .

Various factors, including age, gender, infection severity, local ischemia, diabetes duration, neuropathy, and blood sugar control, are considered potential predictors for DF outcome. However, there remains a lack of complete this study aim to Assessment of predictors of diabetic foot development and outcome in chronic kidney disease patients.

DETAILED DESCRIPTION:
About 537 million adults are living with diabetes mellitus (DM). This number is predicted to rise to 643 million by 2030 . Diabetic foot (DF), being one of the most prevalent, severe, and costly complications of DM. It is primarily characterized by skin infections, ulcers, or destruction of deep tissues below the ankle joint. It is commonly associated with neuropathy or vascular disorders in the lower extremities, and in severe cases, it may involve muscles and bones . Ultimately, 19% to 34% of patients with diabetes will suffer from DF during their lifetimes . Around 20% of DF patients may require lower limb amputations, which can be either minor (below the ankle joint) or major (above the ankle joint), and sometimes both .

Individuals with diabetic neuropathy and Chronic kidney disease (CKD) are 15 times more likely to have a non-traumatic lower extremity amputation compared to those with DM alone . The incidence of DF and its evolution appear to be proportionally related to the stage of CKD . One of the most important causes is vascular calcification, which is common in patients with atherosclerosis, DM, CKD, and elderly .

Various factors, including age, gender, infection severity, local ischemia, diabetes duration, neuropathy, and blood sugar control, are considered potential predictors for DF outcome. However, there remains a lack of complete understanding regarding the most significant factors and their respective impact on the outcome .

ELIGIBILITY:
Inclusion Criteria:

* - Age ≥18 years old.
* TYPE 2 DM with or without DF .
* Patients are at different stages of CKD as defined according to KDIGO (9).

Exclusion Criteria:

* - Patients on dialysis or CKD stage 5 (GFR < 15 ml/min)
* Patients with kidney transplant
* Pregnant patients
* Type 1 DM

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: diabetic nephropathy patients will be divided into two groups ( DF and non-DF groups, 30 patients for each group).
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Ankle brachial index as a predictor for diabetic foot | baseline
  Ankle brachial index is calculated for each leg. The ABI value is determined by taking the higher pressure of the 2 arteries at the ankle, divided by the brachial arterial systolic pressure. In calculating the ABI, the higher of the two brachial systolic pressure measurements is used. In normal individuals, there should be a minimal (less than 10 mm Hg) interarm systolic pressure gradient during a routine examination. A consistent difference in pressure between the arms greater than 10mmHg is suggestive of (and greater than 20mmHg is diagnostic of) subclavian or axillary arterial stenosis, which may be observed in individuals at risk for atherosclerosis

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Abbas ZG, Archibald LK. Challenges for management of the diabetic foot in Africa: doing more with less. Int Wound J. 2007 Dec;4(4):305-13. doi: 10.1111/j.1742-481X.2007.00376.x. Epub 2007 Oct 24. PMID 17961157
- [Result] Levin A, Ahmed SB, Carrero JJ, Foster B, Francis A, Hall RK, Herrington WG, Hill G, Inker LA, Kazancioglu R, Lamb E, Lin P, Madero M, McIntyre N, Morrow K, Roberts G, Sabanayagam D, Schaeffner E, Shlipak M, Shroff R, Tangri N, Thanachayanont T, Ulasi I, Wong G, Yang CW, Zhang L, Robinson KA, Wilson L, Wilson RF, Kasiske BL, Cheung M, Earley A, Stevens PE. Executive summary of the KDIGO 2024 Clinical Practice Guideline for the Evaluation and Management of Chronic Kidney Disease: known knowns and known unknowns. Kidney Int. 2024 Apr;105(4):684-701. doi: 10.1016/j.kint.2023.10.016. PMID 38519239
- [Result] Bonnet JB, Sultan A. Narrative Review of the Relationship Between CKD and Diabetic Foot Ulcer. Kidney Int Rep. 2021 Dec 21;7(3):381-388. doi: 10.1016/j.ekir.2021.12.018. eCollection 2022 Mar. PMID 35257052
- [Result] Gutekunst DJ, Smith KE, Commean PK, Bohnert KL, Prior FW, Sinacore DR. Impact of Charcot neuroarthropathy on metatarsal bone mineral density and geometric strength indices. Bone. 2013 Jan;52(1):407-13. doi: 10.1016/j.bone.2012.10.028. Epub 2012 Oct 29. PMID 23117208